CLINICAL TRIAL: NCT01471249
Title: Quality of Life and Dysphagia Following Palliative Stenting in Esophageal Cancer (CT0023)
Brief Title: Quality of Life and Dysphagia Following Palliative Stenting in Esophageal Cancer
Status: Terminated | Type: Observational
Why Stopped: Insuffisant personnel
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: CE 11.039
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Esophageal Cancer
Keywords: esophageal stenting; palliative; dysphagia
MeSH Terms: conditions — Esophageal Neoplasms; Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study consists of a prospective clinical trial which aims to evaluate the impact of stent insertion for palliation of malignant dysphagia. The main goal being to examine the number of days required following stenting in order to have significant improvement in dysphagia and the length of time that this baseline is maintained. Approximately 100 patients will be prospectively enrolled in this study.

Patients with end stage inoperable esophageal cancer deemed candidates for intraluminal esophageal palliative stent insertion will be prospectively enrolled into the study. Patients with esophageal obstruction or stricture due to other benign causes, tumors obstructing the cervical esophagus, as well as patients with airway-esophageal fistulas will be excluded from the study.

The investigators plan to evaluate the efficacy of intra-esophageal stent insertion to improve malignant dysphagia as a main factor affecting the quality of life in these patients.

DETAILED DESCRIPTION:
Esophageal cancer is one of the 10 most frequent cancers in the world. The incidence of esophageal cancer is rapidly increasing and is doing so at a more rapid rate than any other cancer in the western world. The annual incidence reported in western countries is 3 per 100,000. In central China it has been reported to be as high as 140 per 100,000 in Linxian Province in central China.

Esophageal cancer remains one of the most lethal of all malignancies. Once a diagnosis is established, the prognosis is poor, with a 5-year survival rate of less than 10%. Despite advances in therapy, more than 50% of patients have incurable disease at the time of presentation and only one third of patients with localized disease experience long term survival.

By the appearance of dysphagia and by the time of diagnosis, most patients are not candidates for esophagectomy because symptoms are not present until at least 50% of the circumference of the oesophagus is involved. Distant metastasis will usually be established by this time.

The symptoms of dysphagia and weight loss that are commonly experienced have a significant impact on quality of life for these patients. This makes palliative endoluminal stenting an attractive option. The mainstay of treatment is the palliation of dysphagia resulting from malignant stenosis and intraluminal tumor growth.

A number of palliative therapies are available to the treating physician. The options for treating dysphagia that is caused by advanced, unresectable esophageal cancer include: stenting, photodynamic therapy (PDT), thermal laser ablation, external beam radiation and brachytherapy.

Brachytherapy offers safe palliation for malignant dysphagia over a relatively long period. The results of brachytherapy are comparable to the other palliative methods. Increased effectiveness and more symptomatic improvements have been reported with the combination of external beam radiation with high dose brachytherapy. The combination was well tolerated and relatively safe. Despite relatively safe, perforation and stricture formation are complications for brachytherapy with or without external beam radiation. Furthermore, brachytherapy has fallen out of favour in most centers due to the time to amelioration of symptoms and the required multiple hospital visits for repeated procedures.

Photodynamic therapy (PDT) utilizes a photosensitizing agent, light and oxygen to endoscopically ablate cancer cells. PDT has been suggested and evaluated for the treatment of high grade esophageal dysplasia and intramucosal adenocarcinoma arising within Barrett's oesophagus. Ablation with PDT has been effective for end stage esophageal cancer palliation and improving malignant dysphagia. Esophagitis, photoreactions, perforation, and strictures requiring dilatation are still the main complications for PDT and have been the reason for its disappearance from clinical practise.

Laser and thermal ablation are commonly used methods for esophageal cancer palliation. Despite relatively good results, perforation, and the necessity for re-intervention are the main concern that limit their use for most end stage esophageal cancer patients.

Intra luminal esophageal stenting is widely used as an effective method for esophageal cancer palliation. Esophageal stent insertion proved to be an effective method for palliation of malignant dysphagia. It is a relatively safe procedure with a low rate of serious complications. In a report of 127 stent placements in 100 patients, immediate relief of dysphagia was observed with the stent insertion in 85% of patients. Adding to its proven efficacy for treatment of dysphagia, stenting was proven to offer palliation with longer interventional free periods than any other methods of palliation. Over the past decade, advances in expandable stent technology have led to smaller, more flexible delivery systems that are easier to manipulate than the original plastic stents. These attributes permit successful deployment without exposing patients to the risks of aggressive mechanical dilatation.

Stent insertion is also the only effective method for palliation of esophageal cancer with extrinsic compression (metastatic mediastinal lymph nodes) causing dysphagia. Stenting also plays an important role in treatment of patients with airway - esophageal fistulas.

This study consists of a prospective clinical trial which aims to evaluate the impact of stent insertion for palliation of malignant dysphagia. The main goal being to examine the number of days required following stenting in order to have significant improvement in dysphagia and the length of time that this baseline is maintained.

Hypothesis:

Intraluminal esophageal stenting improves malignant dysphagia and quality of life almost immediately after stent insertion and this effect is maintained in the short and medium term in inoperable esophageal cancer patients.

Objectives:

* To assess the effectiveness of esophageal stenting in improving malignant dysphagia and assess the time period relating to this improvement
* To assess the effectiveness of esophageal stenting in improving quality and assess the time period relating to this improvement

Study design:

Prospective non-interventional clinical trial.

Methods:

Patients with malignant dysphagia who are scheduled for palliative endoluminal esophageal stenting will be prospectively enrolled into the trial. All patients eligible for the study will be consented by study investigators in the outpatient clinic prior to their procedure. Study investigators will administer the questionnaires following consent.

Patients will undergo the standard endoscopic intervention of intraluminal esophageal stent insertion.

Assessment of dysphagia score will be performed immediately prior to the procedure, after the procedure (day 0), as well as days 1 to 7, then every week for 4 weeks post procedure.

Questionnaires performed by study investigators will take place in either the clinic before the operation or in Notre-Dame hospital during hospital stay. Later questionnaires will be performed by telephone interview.

Analysis will aim to compare dysphagia and quality of life scores between baseline (pre-procedure) values and post-procedural values. The time to achieve a steady state will also be assessed. Maintenance of improved quality of life and of low dysphagia score will also be assessed. Secondary outcome will be a survival analysis based on stage.

ELIGIBILITY:
Inclusion Criteria:

* All patients with end stage inoperable esophageal cancer deemed candidates for intraluminal esophageal palliative stent insertions.

Exclusion Criteria:

* Inability to consent for the study.
* Patients less than 18 years old.
* Patients with other benign causes of dysphagia and esophageal obstruction or stenosis.
* Patients with malignant or benign airway - esophageal fistulas.
* Patients with cervical esophageal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients referred to the thoracic clinic or in-patient
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2011-06; Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
improvement of dysphagia post stenting | 3 months
  To assess the effectiveness of esophageal stenting in improving malignant dysphagia and assess the time period relating to this improvement

SECONDARY OUTCOMES:
Quality of life post stenting | 3 months
  To assess the effectiveness of esophageal stenting in improving quality of life and assess the time period relating to this improvement

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, PhD, Principal Investigator — CHUM-Centre Universitaire de Montreal
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada